CLINICAL TRIAL: NCT07151859
Title: A Pre-market, Two-stages, Monocentric, Interventional, Single-arm, Clinical Investigation to Evaluate the Safety and the Performance of PN30 (RDM16) for the Improvement of Skin Hydration
Brief Title: Clinical Investigation on a Polynucleotide-based Device Used to Improve Skin Hydration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mastelli S.r.l (Industry)
Collaborators: 1Med (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-PN30-2024
Record Dates: First submitted 2025-08-07; First posted 2025-09-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Aesthetic Improvement of the Skin; Skin Hydration in Healthy Volunteers; Skin Elasticity; Skin Turgor; Subject Satisfaction
Keywords: aesthetic; Polynucleotides; PN HPT; skin; skin quality; skin elasticity; skin turgor; skin hydration; face; neck; décolleté
MeSH Terms: conditions — Facies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Device: PN30 (RDM16)

INTERVENTIONS:
Device: PN30 (RDM16) — PN30 is a viscoelastic, sterile gel, in a disposable prefilled syringe for intradermal infiltration.PN30 contains polynucleotides (3%). The polynucleotides contained in the device are substances of natural, fish-derived origin, highly purified.

SUMMARY:
Adequate skin hydration is critical for maintaining healthy skin. Moreover, dehydration, together with reduction in cell renewal, loss of radiance, elasticity and firmness, is involved in skin aging. Injectable anti-aging products have been widely used for aesthetic improvement of the skin.

In recent years, new filler products made from High Purification Technology Polynucleotides (PN HPTTM) have been developed and are now being used in Europe. PN HPTTM has a consolidated utilization in the aesthetic field and recently, specific guidelines in their utilization have been implemented. Polynucleotides (PNs) are polymeric chains formed by purines, pyrimidines, deoxyribonucleotides, and deoxyribonucleosides that can be found in cells throughout the human body. PNs have viscoelastic properties and the capability to bind, reorganize and orientate a high concentration of water molecules, creating 3D gel that undergoes an enzymatic cleavage.

On this basis, polynucleotide-containing products act as short-time temporary fillers to produce a volumizing effect and exert a lubricant and moisturizing action, due to the high concentration of water molecules. Moreover, they maintain for a long time the moisturizing and viscoelastic effect.

A recent report which summarizes the findings and recommendations issued from the Italian Scientific Board of aesthetic physicians, supports the use of PN-HPT.

In this context, the Sponsor has developed PN30, a soft-tissue filler containing PN-HPT (at a concentration of 30 mg/ mL) as functional ingredients which help improve skin turgor and elasticity due to their moisturizing and viscoelastic properties.

PN30 is a new device with no history of marketing but based on a similar product CE marked developed and sold by the Manufacturer with less amount of PN (2%). Therefore, the aim of this pre-market, twostages, monocentric, interventional, single-arm, clinical investigation is to evaluate the safety and the performance of PN30 (RDM16) for the improvement of skin hydration. The clinical investigation is planned as an adaptative two-stages study.

The planned procedures will be the same for both stages. The primary objective/endpoint of STAGE I will be to evaluate the safety, while the primary objective/endpoint of STAGE II will be to evaluate the performance of the device.

ELIGIBILITY:
Inclusion Criteria:

1. Subject Informed consent form (ICF) signed;
2. Female and male Subjects aged 18-70 years;
3. Subjects desiring improvement of skin hydration in maximum 1 area of the face or desiring improvement of skin hydration of neck or décolleté.
4. Healthy skin;
5. Willingness to discontinue all dermatological treatment and procedures during the study;
6. Willingness to follow all study procedures, including attending all site visits, tests and examinations;
7. Agreeing to present at each study visit without face/neck/décolleté cosmetics;
8. Accepting to not change their habits regarding food, physical activity, face/neck/décolleté cosmetics and cleansing products;
9. Willingness to follow indications to avoid make-up in the 12 hours following the injection treatment and to avoid any prolonged exposure to the sun, UV rays and temperatures below 0°C, as well as any sauna or hammam sessions at least until the wheals have been fully reabsorbed;
10. Skin phototype I-IV according to Fitzpatrick's classification.

Exclusion Criteria:

1. Other - different - clinical conditions of the skin (i.e. rosacea, psoriasis, vitiligo, active eczema, severe scleroderma, severe acne and diagnosticated cancer with/without ongoing antitumor therapy);
2. Infectious or inflammatory processes near the area of intervention;
3. Presence of cutaneous disease on the tested area, as malformations and recurrent facial/labial herpes;
4. Presence of tendon, bone or muscular implants near the area of intervention;
5. Ongoing cutaneous allergies;
6. Allergy or contraindications to device components;
7. Concomitant intake of anticoagulant or antiplatelet medications;
8. Subjects who have not followed a washout period of 2 weeks from topical corticosteroids, antibiotics, benzoyl-peroxide, azelaic acid, hydroxy acids, topical retinoids;
9. Immune system illnesses/disease;
10. Uncontrolled diabetes mellitus or uncontrolled systemic diseases (endocrine, hepatic renal, cardiac, pulmonary, neurological disorder);
11. Treatment with substances which act on blood fluidity (eg. Aspirin, NSAIDs, Vitamin E), or drugs able to influence the test results in the investigator opinion, within 5 days prior to study inclusion;
12. Known drug and/or alcohol abuse;
13. Mental incapacity that precludes adequate understanding or cooperation;
14. Any previous permanent and non-permanent cutaneous treatment for aesthetic correction (biomaterial implant, lifting, laser, botulinum toxin injections, chemical peeling, fillers) of the treated area within 6 months prior to study inclusion;
15. Pregnancy or breastfeeding;
16. Participation in another investigational study within 1 month prior to study inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Stage I - Skin examination (through evaluation of possible cutaneous reactions) | From enrollment to the end of study at 12 weeks ± 7 days after last treatment
Stage I - Device deficiencies monitoring | At baseline (first injection) and 5 weeks ± 7 days from baseline (second and last injection)
  A device deficiency (DD) is any inadequacy in the identity, quality, durability, reliability, safety or performance of an investigational device, including malfunction, use errors or inadequacy in information supplied by the manufacturer. This definition includes device deficiencies related to the investigational medical device. The rate of DD will be assessed and counted by the investigator at baseline (Visit 0), at Visit 1 and at Visit 2.
Stage I - Adverse events, serious adverse events and concomitant medications monitoring. | From enrollment to the end of study at 12 weeks ± 7 days after last treatment
  Adverse events, serious adverse events and concomitant medications will be monitored during the entire study duration. Subjects will receive a diary to record any deviation from the normal health status as well as any concomitant medication taken.
Stage II - Aesthetic evaluation of the skin through the change in Global Aesthetic Improvement Scale (GAIS) completed per each area treated by the Investigator | 10 weeks from the last treatment
  To evaluate the performance of PN30 for the aesthetic improvement of the skin after 10 weeks from the last treatment, the change in Global Aesthetic Improvement Scale (GAIS, rated on a 5-point scale (1= very much/extremely improved; 2= much improved; 3= improved; 4= no change; 5= worse)) from V2 to baseline (pre-treatment) will be assessed. The GAIS will be completed per each area treated by the Investigator. The pre-treatment GAIS score (at baseline/V0) will be "4" for each area treated for all subjects enrolled.

SECONDARY OUTCOMES:
Stage I and Stage II - Aesthetic evaluation of the skin through the change in Global Aesthetic Improvement Scale (GAIS) completed per each area treated by the Investigator | From enrollment to the end of study at 12 weeks ± 7 days after last treatment
  To evaluate the performance of PN30 for the aesthetic improvement of the skin at each visit, the change in Global Aesthetic Improvement Scale (GAIS, rated on a 5-point scale (1= very much/extremely improved; 2= much improved; 3= improved; 4= no change; 5= worse)) will be assessed. The GAIS will be completed per each area treated by the Investigator. The pre-treatment GAIS score (at baseline/V0) will be "4" for each area treated for all subjects enrolled.
Stage I and Stage II - Evaluation the performance of PN30 on skin hydration at each visit through the MoistureMeterEpiD | From enrollment to the end of study at 12 weeks ± 7 days after last treatment
  The MoistureMeterEpiD (Delfin Technology, Finland) generates a high frequency (300 MHz), low power electromagnetic (EM) wave which the tissue is exposed to. The reflected EM wave is registered, and the obtained value is a dielectric constant (TDC), which is proportional to the water content of the measured tissue. The value increases with increasing water content. The dielectric constant is converted to water percentage (0-100%).
Stage I and Stage II - Evaluation the performance of PN30 on skin elasticity at each visit through the ElastiMeter | From enrollment to the end of study at 12 weeks ± 7 days after last treatment
  The ElastiMeter (Delfin Technology, Finland) comprises a reference plate with an indenter located at the centre. As the instrument is pressed briefly against the skin, a constant deformation to the skin surface is produced without altering the skin structure. A sensor measures the force required to produce the deformation from which the instant skin elasticity can be determined. The ElastiMeter measures skin elasticity in N/m.
Stage I and Stage II - Evaluation of the performance of PN30 on skin turgor at each visit through a 5-point Likert scale assessed by the Investigator | From enrollment to the end of study at 12 weeks ± 7 days after last treatment
  A 5-point Likert scale is a survey tool with five response options designed to measure the opinions, including two negative options, one neutral option, and two positive options.
Stage I and Stage II - Injection pain intensity through the Numerical Rating Scale (NRS) | At baseline (first injection) and 5 weeks ± 7 days from baseline (second and last injection)
  The NRS consists of an 11-point scale from 0 to 10, where 0 means "no pain" and 10 represents "worst imaginable pain". The NRS can be administered verbally soon after the injection or by telephone after the injection, if anesthesia is performed. In this case, the Investigator should wait until the effect of anesthesia is resolved before asking the Subject the numerical value that best describes her/his pain intensity.
Stage I and Stage II - Evaluation of the subject satisfaction through a 5-point Likert scale | 10 weeks ± 7 days after last treatment and 12 weeks ± 7 days after last treatment (End Of Study)
  To evaluate subject satisfaction with PN30, a 5-Likert scale, from 1 to 5 indicating how satisfied is the patient (1 - Extremely dissatisfied, 5 - Extremely satisfied), will be used at Visit 2 and at End of study (Visit 3)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria "Federico II", Napoli, Italy, Italy